CLINICAL TRIAL: NCT05895916
Title: Extreme Exercise and Energy Expenditure (4E) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Responsible Party: Principal Investigator, Natalie Alméras, Principal Investigator, Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 4E study
Record Dates: First submitted 2023-05-17; First posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-05

CONDITIONS: Cardiovascular Diseases; Obesity, Visceral; Liver Fat; Metabolic Syndrome; Lifestyle
Keywords: cardiac fat; cardiometabolic health; cardiorespiratory fitness; ectopic fat; energy balance; exercise; liver fat; obesity; physical activity; visceral adipose tissue
MeSH Terms: conditions — Cardiovascular Diseases; Obesity, Abdominal; Fatty Liver; Metabolic Syndrome; Motor Activity; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Extreme exercise group (Experimental): 1,144 km of road cycling on seven consecutive days
  Interventions: Behavioral: High-volume road cycling

INTERVENTIONS:
Behavioral: High-volume road cycling — 1,144 km of road cycling performed on seven consecutive days with an increase in energy intake to maintain a stable body weight

SUMMARY:
The goal of this clinical trial is to provide evidence, through an extreme exercise prescription (1,144 km of road cycling on seven consecutive days), that weight loss is not the appropriate outcome to evaluate the effects of exercise on abdominal adiposity and ectopic fat depots (e.g. liver fat and epi/pericardial fat) in eleven recreational middle-aged male cyclists (aged 50 to 66 years) without symptoms of cardiovascular disease. The main questions it aims to answer are:

* If energy intake is substantially increased to compensate energy expenditure and prevent weight loss following an extreme exercise prescription, will significant changes in body composition and body fat distribution be observed?
* Will these changes translate into improvements in the cardiometabolic health profile even in the absence of weight loss?

Participants will be asked to partake in several evaluations: fasting plasma lipoprotein-lipid profile and inflammation markers, glycated hemoglobin, cardiorespiratory fitness, submaximal exercise test including measurement of energy expenditure, resting and exercise blood pressure and heart rate, evaluation of regional adiposity, liver fat content, epi/pericardial fat, nutritional quality, and level of physical activity. After baseline evaluations, participants will be asked to alternately bike 208 km and 104 km per day on a pre-specified course for seven consecutive days. They will be accompanied during each of the seven bike rides by research professionals in a recreational vehicle. Participants' weight, body composition and waist circumference will be measured under standardized conditions in the morning after an overnight fast and after the exercise. Their heart rate will be continuously monitored, and participants will wear accelerometers to estimate their daily exercise-related energy expenditure. Foods and fluids will be provided to participants and recorded. At the end of the 1,144 km/ 7-days bike ride, baseline evaluations will be repeated with the exception of the maximal exercise treadmill test, nutritional quality, and level of physical activity. To facilitate the conduct of the protocol, the eleven participants will be evaluated and followed in two distinct groups.

DETAILED DESCRIPTION:
Although there is robust evidence that a physically active lifestyle including regular leisure time physical activity and exercise (>150 min per week of moderate to vigorous exercise per week) is associated with a reduced mortality risk and improved cardiometabolic health, some scientists have promoted the notion (which has certainly been taken up by the lay press) that if one wants to lose weight, focus should be placed on caloric restriction rather than on exercise. Several academic debates have been held on this issue which have left some health professionals and the public confused and perplexed.

The investigators' research group has been active in this area on several fronts. First, the investigators have pioneered the notion that in cardiovascular and "metabolic" medicine, the health risk of overweight and obesity was not appropriately assessed by an index based on body weight (body mass index, which is expressed in kg/m^2). For instance, using imaging technology (computed tomography), the investigators were among the first, more than 30 years ago, to begin to extensively study regional body fat distribution, showing that excess visceral adipose tissue accumulation was more closely related to an atherogenic and diabetogenic cardiometabolic risk profile than excess body weight or total body fat. As sedentary individuals with a diet of poor nutritional value (rich in processed fat and added sugar - promoting preferential visceral fat deposition) are also often characterized by a lower muscle mass and by high levels of abdominal visceral fat, several lifestyle intervention studies that the investigators and others have conducted in sedentary males with visceral obesity have shown that with regular exercise, one could lose visceral adipose tissue while gaining muscle mass, which would lead to trivial or sometimes no changes in body weight. Thus, if body composition is altered by an energy deficit produced by regular exercise, the investigators have proposed that weight loss may sometime be misleading as an outcome as it may not always reflect favorable changes in body composition (muscle mass increasing) and in visceral adiposity and levels of ectopic fat (decreasing). On that basis, the investigators have proposed that changes in waist circumference could be more useful than body weight loss in the evaluation of the benefits of a lifestyle modification program involving regular endurance exercise such as brisk walking, jogging, or biking. For instance, the investigators have previously reported that waist circumference was rather sensitive to lifestyle changes involving regular physical activity/exercise. Accordingly, lifestyle intervention studies have shown that a reduction of 4 cm in waist girth was predictive of a 58% reduction in the risk of developing type 2 diabetes among individuals who were initially characterized by abdominal obesity and glucose intolerance.

Thus, there is a need to propose a paradigm shift among health professionals to evaluate the impact of lifestyle intervention programs involving physical activity/exercise in high-risk overweight obese individuals with visceral obesity: Weight loss is no longer the optimal or most clinically relevant outcome - losses of visceral adiposity and ectopic fat may be more relevant clinically.

In 2015, a member of the investigators' team was asked to write an editorial on a spectacular study which provided very relevant data to the debate about diet vs. exercise and weight loss. In that impressive exercise study, recreational middle-aged cyclists were required to bike 2,700 km over 14 days and asked to try to match their energy intake to their very large energy expenditure, the objective being not to lose weight over the course of the intervention. Thus, the daily exercise "prescription" was huge as the authors wanted to test the ability of these elderly and fit recreational cyclists to match their energy intake to their energy expenditure. The most striking and important finding of this unusual study is that despite the huge energy expenditure associated with the 2,700 km bike expedition, participants did not lose weight. However, such lack of change in body weight was completely misleading in terms of energy balance and changes in body composition. Indeed, the cyclists lost 2.2 kg of body fat while gaining 2.5 kg of fat-free mass, a remarkable finding considering that such changes were observed over a period of only two weeks.

Results of this study provide additional evidence that body weight is a poor outcome to assess the effect of a physical activity/exercise program. In the investigators' previously published exercise training studies, a common observation has been the disconnect between changes in body weight and changes in body composition, the latter being sometime observed even in the absence of weight loss. As weight poorly tracks changes in body composition induced by exercise, no wonder why exercise is indeed perceived as not being helpful to lose weight by some health professionals. The investigators propose that body weight is a misleading outcome when comes the time to evaluate the clinical benefits of exercise in individuals with overweight/obese.

One remaining and clinically important issue remains to be addressed regarding the effects of a large volume of exercise not inducing weight loss: to what extent substantial changes in visceral/ectopic fat could have been observed had imaging data been available? In addition, it would have been interesting for the 2,700 km bike intervention study to report changes in waist circumference, this metric being more sensitive to regular exercise than body weight. In the investigators' previous intervention studies, it has been their experience to find participants losing quite a bit of visceral fat and dropping their waistline by several centimeters, while not losing any body weight.

Thus, on the basis of the above observations, the investigators put forward the hypotheses that:

1. a very large volume of exercise (1,144 km of bicycle performed for 7 consecutive days) will induce major changes in body composition and in levels of visceral adipose tissue/ectopic fat in a sample of middle-aged recreational cyclists who will be asked to match their energy intake to their very large energy expenditure during the course of the one-week extreme exercise intervention. Thus, in a study where, by design, no weight loss is planned nor wanted, the investigators expect to see major changes in body composition (slight increase in muscle mass and substantial reductions in the size of visceral adipose tissue and ectopic fat depots);
2. changes in levels of visceral adipose tissue and ectopic fat will be better reflected by changes in waist circumference - which should decrease in the absence of body weight loss.

The investigators recognize that this is an extreme exercise prescription that has little relevance to public health. However, results of this study will be very important in shedding light on the importance of shifting our attention from body weight loss to other, more clinically relevant fat depots. Thus, the purpose of the study is to provide evidence, through an extreme exercise prescription, that weight loss is not the appropriate outcome to evaluate the effects of exercise on visceral adiposity and ectopic fat depots (e.g. liver fat and epi/pericardial fat) which will likely be mobilized to a very significant extent in only one week.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Between the ages of 50 and 66 years
* Asymptomatic for cardiovascular disease
* Reporting at least 5,000 km per year of road cycling at an average pace of about 30 km/h

Exclusion Criteria:

* Retired competitive athletes/competitive athletes
* Undergoing hormonal or corticosteroid therapy
* Presenting a cancer not in remission
* Presenting an absolute contraindication to MRI
* Presenting an absolute contraindication to maximal cardiopulmonary exercise testing

Ages: 50 Years to 66 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2019-08-13 (Actual); Study Completion 2019-08-13 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in body weight assessed by direct segmental multi-frequency bioimpedance analysis following the extreme exercise prescription | Before and the day (or next day) following the extreme exercise prescription
  Changes in body weight in kilograms
Changes from baseline in fat mass assessed by direct segmental multi-frequency bioimpedance analysis following the extreme exercise prescription | Before and the day (or next day) following the extreme exercise prescription
  Changes in fat mass in kilograms
Changes from baseline in fat-free mass assessed by direct segmental multi-frequency bioimpedance analysis following the extreme exercise prescription | Before and the day (or next day) following the extreme exercise prescription
  Changes in fat-free mass in kilograms
Changes from baseline in body water assessed by direct segmental multi-frequency bioimpedance analysis following the extreme exercise prescription | Before and the day (or next day) following the extreme exercise prescription
  Changes in body water in kilograms
Changes from baseline in waist circumference assessed using a standardized measuring tape following the extreme exercise prescription | Before and the day (or next day) following the extreme exercise prescription
  Changes in waist circumference in centimeters
Changes from baseline in visceral adipose tissue assessed using magnetic resonance imaging following the extreme exercise prescription | Before and the day (or next day) following the extreme exercise prescription
  Changes in visceral adipose tissue in milliliters
Changes from baseline in subcutaneous adipose tissue assessed using magnetic resonance imaging following the extreme exercise prescription | Before and the day (or next day) following the extreme exercise prescription
  Changes in subcutaneous adipose tissue in milliliters
Changes from baseline in epicardial adipose tissue assessed using magnetic resonance imaging following the extreme exercise prescription | Before and the day (or next day) following the extreme exercise prescription
  Changes in epicardial adipose tissue in milliliters
Changes from baseline in pericardial adipose tissue assessed using magnetic resonance imaging following the extreme exercise prescription | Before and the day (or next day) following the extreme exercise prescription
  Changes in pericardial adipose tissue in milliliters
Changes from baseline in liver fat content assessed using magnetic resonance imaging with spectroscopy following the extreme exercise prescription | Before and the day (or next day) following the extreme exercise prescription
  Changes in liver fat content in percentage

SECONDARY OUTCOMES:
Changes from baseline in fasting total cholesterol following the extreme exercise prescription | Before and the day (or next day) following the extreme exercise prescription
  Changes in fasting total cholesterol in millimoles per liter
Changes from baseline in fasting LDL cholesterol following the extreme exercise prescription | Before and the day (or next day) following the extreme exercise prescription
  Changes in fasting LDL cholesterol in millimoles per liter
Changes from baseline in fasting HDL cholesterol following the extreme exercise prescription | Before and the day (or next day) following the extreme exercise prescription
  Changes in fasting HDL cholesterol in millimoles per liter
Changes from baseline in fasting plasma triglycerides following the extreme exercise prescription | Before and the day (or next day) following the extreme exercise prescription
  Changes in fasting plasma triglycerides in millimoles per liter
Changes from baseline in fasting glycated hemoglobin following the extreme exercise prescription | Before and the day (or next day) following the extreme exercise prescription
  Changes in fasting glycated hemoglobin in percentage
Changes from baseline in fasting apolipoprotein A1 following the extreme exercise prescription | Before and the day (or next day) following the extreme exercise prescription
  Changes in fasting apolipoprotein A1 in grams per liter
Changes from baseline in fasting apolipoprotein B following the extreme exercise prescription | Before and the day (or next day) following the extreme exercise prescription
  Changes in fasting apolipoprotein B in grams per liter
Changes from baseline in fasting adiponectin following the extreme exercise prescription | Before and the day (or next day) following the extreme exercise prescription
  Changes in fasting adiponectin in micrograms per milliliter
Changes from baseline in fasting leptin following the extreme exercise prescription | Before and the day (or next day) following the extreme exercise prescription
  Changes in fasting leptin in nanograms per milliliter
Changes from baseline in fasting C-reactive protein following the extreme exercise prescription | Before and the day (or next day) following the extreme exercise prescription
  Changes in fasting C-reactive protein in milligrams per liter
Changes from baseline in fasting interleukin-6 following the extreme exercise prescription | Before and the day (or next day) following the extreme exercise prescription
  Changes in fasting interleukin-6 in picograms per milliliter
Changes from baseline in fasting tumor necrosis factor alpha following the extreme exercise prescription | Before and the day (or next day) following the extreme exercise prescription
  Changes in fasting tumor necrosis factor alpha in picograms per milliliter
Changes from baseline in resting systolic blood pressure following the extreme exercise prescription | Before and the day (or next day) following the extreme exercise prescription
  Changes in resting systolic blood pressure in millimeters of mercury
Changes from baseline in resting diastolic blood pressure following the extreme exercise prescription | Before and the day (or next day) following the extreme exercise prescription
  Changes in resting diastolic blood pressure in millimeters of mercury

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Alméras, Ph.D., Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec - Université Laval, Québec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kraus WE, Bittner V, Appel L, Blair SN, Church T, Despres JP, Franklin BA, Miller TD, Pate RR, Taylor-Piliae RE, Vafiadis DK, Whitsel L; American Heart Association Physical Activity Committee of the Council on Lifestyle and Metabolic Health, Council on Clinical Cardiology, Council on Hypertension, and Council on Cardiovascular and Stroke Nursing. The National Physical Activity Plan: a call to action from the American Heart Association: a science advisory from the American Heart Association. Circulation. 2015 May 26;131(21):1932-40. doi: 10.1161/CIR.0000000000000203. Epub 2015 Apr 27. No abstract available. PMID 25918126
- [Background] Luke A, Cooper RS. Physical activity does not influence obesity risk: time to clarify the public health message. Int J Epidemiol. 2013 Dec;42(6):1831-6. doi: 10.1093/ije/dyt159. No abstract available. PMID 24415616
- [Background] Malhotra A, Noakes T, Phinney S. It is time to bust the myth of physical inactivity and obesity: you cannot outrun a bad diet. Br J Sports Med. 2015 Aug;49(15):967-8. doi: 10.1136/bjsports-2015-094911. Epub 2015 Apr 22. No abstract available. PMID 25904145
- [Background] Blair SN, Archer E, Hand GA. Commentary: Luke and Cooper are wrong: physical activity has a crucial role in weight management and determinants of obesity. Int J Epidemiol. 2013 Dec;42(6):1836-8. doi: 10.1093/ije/dyt160. No abstract available. PMID 24415617
- [Background] Blair SN. Physical inactivity and obesity is not a myth: Dr. Steven Blair comments on Dr. Aseem Malhotra's editorial. Br J Sports Med. 2015 Aug;49(15):968-9. doi: 10.1136/bjsports-2015-094989. Epub 2015 Jun 10. No abstract available. PMID 26062953
- [Background] Despres JP, Moorjani S, Lupien PJ, Tremblay A, Nadeau A, Bouchard C. Regional distribution of body fat, plasma lipoproteins, and cardiovascular disease. Arteriosclerosis. 1990 Jul-Aug;10(4):497-511. doi: 10.1161/01.atv.10.4.497. PMID 2196040
- [Background] Despres JP, Lemieux I, Bergeron J, Pibarot P, Mathieu P, Larose E, Rodes-Cabau J, Bertrand OF, Poirier P. Abdominal obesity and the metabolic syndrome: contribution to global cardiometabolic risk. Arterioscler Thromb Vasc Biol. 2008 Jun;28(6):1039-49. doi: 10.1161/ATVBAHA.107.159228. Epub 2008 Mar 20. PMID 18356555
- [Background] Despres JP. Body fat distribution and risk of cardiovascular disease: an update. Circulation. 2012 Sep 4;126(10):1301-13. doi: 10.1161/CIRCULATIONAHA.111.067264. No abstract available. PMID 22949540
- [Background] Borel AL, Nazare JA, Smith J, Almeras N, Tremblay A, Bergeron J, Poirier P, Despres JP. Visceral and not subcutaneous abdominal adiposity reduction drives the benefits of a 1-year lifestyle modification program. Obesity (Silver Spring). 2012 Jun;20(6):1223-33. doi: 10.1038/oby.2011.396. Epub 2012 Jan 19. PMID 22262155
- [Background] Ross R, Dagnone D, Jones PJ, Smith H, Paddags A, Hudson R, Janssen I. Reduction in obesity and related comorbid conditions after diet-induced weight loss or exercise-induced weight loss in men. A randomized, controlled trial. Ann Intern Med. 2000 Jul 18;133(2):92-103. doi: 10.7326/0003-4819-133-2-200007180-00008. PMID 10896648
- [Background] Despres JP. Obesity and cardiovascular disease: weight loss is not the only target. Can J Cardiol. 2015 Feb;31(2):216-22. doi: 10.1016/j.cjca.2014.12.009. Epub 2014 Dec 11. PMID 25661557
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Tuomilehto J, Lindstrom J, Eriksson JG, Valle TT, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Laakso M, Louheranta A, Rastas M, Salminen V, Uusitupa M; Finnish Diabetes Prevention Study Group. Prevention of type 2 diabetes mellitus by changes in lifestyle among subjects with impaired glucose tolerance. N Engl J Med. 2001 May 3;344(18):1343-50. doi: 10.1056/NEJM200105033441801. PMID 11333990
- [Background] Despres JP. Exercise and energy balance: going to extremes to show that body weight is not the best outcome. Am J Clin Nutr. 2015 Dec;102(6):1303-4. doi: 10.3945/ajcn.115.124560. Epub 2015 Nov 11. No abstract available. PMID 26561630
- [Background] Rosenkilde M, Morville T, Andersen PR, Kjaer K, Rasmusen H, Holst JJ, Dela F, Westerterp K, Sjodin A, Helge JW. Inability to match energy intake with energy expenditure at sustained near-maximal rates of energy expenditure in older men during a 14-d cycling expedition. Am J Clin Nutr. 2015 Dec;102(6):1398-405. doi: 10.3945/ajcn.115.109918. Epub 2015 Oct 21. PMID 26490491
- [Background] Iacobellis G, Ribaudo MC, Assael F, Vecci E, Tiberti C, Zappaterreno A, Di Mario U, Leonetti F. Echocardiographic epicardial adipose tissue is related to anthropometric and clinical parameters of metabolic syndrome: a new indicator of cardiovascular risk. J Clin Endocrinol Metab. 2003 Nov;88(11):5163-8. doi: 10.1210/jc.2003-030698. PMID 14602744
- [Background] Iacobellis G, Leonetti F. Epicardial adipose tissue and insulin resistance in obese subjects. J Clin Endocrinol Metab. 2005 Nov;90(11):6300-2. doi: 10.1210/jc.2005-1087. Epub 2005 Aug 9. PMID 16091479
- [Background] Rosito GA, Massaro JM, Hoffmann U, Ruberg FL, Mahabadi AA, Vasan RS, O'Donnell CJ, Fox CS. Pericardial fat, visceral abdominal fat, cardiovascular disease risk factors, and vascular calcification in a community-based sample: the Framingham Heart Study. Circulation. 2008 Feb 5;117(5):605-13. doi: 10.1161/CIRCULATIONAHA.107.743062. Epub 2008 Jan 22. PMID 18212276
- [Background] De Larochelliere E, Cote J, Gilbert G, Bibeau K, Ross MK, Dion-Roy V, Pibarot P, Despres JP, Larose E. Visceral/epicardial adiposity in nonobese and apparently healthy young adults: association with the cardiometabolic profile. Atherosclerosis. 2014 May;234(1):23-9. doi: 10.1016/j.atherosclerosis.2014.01.053. Epub 2014 Feb 7. PMID 24589564
- [Background] Almeras N, Mimeault N, Serresse O, Boulay MR, Tremblay A. Non-exercise daily energy expenditure and physical activity pattern in male endurance athletes. Eur J Appl Physiol Occup Physiol. 1991;63(3-4):184-7. doi: 10.1007/BF00233845. PMID 1761005

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/16/NCT05895916/Prot_SAP_000.pdf